CLINICAL TRIAL: NCT06196450
Title: Ability of the Probiotic Vivomixx to Improve Environmental Enteropathy in Pregnant Women: a Proof of Concept Trial in Bangladesh, Pakistan, Senegal and Zambia
Brief Title: Maternal Probiotic Intervention to Improve Gut Health
Acronym: MPIGH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PR-22084
Record Dates: First submitted 2023-06-05; First posted 2024-01-09 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Environmental Enteric Dysfunction; Gut Microbiota Dysbiosis
Keywords: probiotic; gut health; GWG; fetal growth; perinatal outcome

STUDY DESIGN:
Intervention Model Description: Multi-site phase II randomised controlled trial (Proof of concept study)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Vivomixx and Placebo (Crystalline maltose)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Vivomixx also known as VSL#3, Powder (in sachets), weight 4.4g, 450 X 10^9 cfu of probiotic bacteria per sachet, dose 1 sachet daily for 56 days
  Interventions: Dietary Supplement: Vivomixx
- Placebo arm (Placebo Comparator): Microcrystalline maltose, Powder (in sachets), weight 4.4g, dose 1 sachet daily for 56 days
  Interventions: Dietary Supplement: Microcrystalline maltose

INTERVENTIONS:
Dietary Supplement: Vivomixx — Vivomixx is a commercially available probiotic mixture consisting of eight probiotic lactic acid bacteria and Bifidobacteria including Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus casei, Lactobacillus delbrueckii subspecies bulgaricus, Streptococcus salivarius subspecies thermophiles, Bifidobacterium breve, Bifidobacterium longum, and Bifidobacterium infantis.
  Arms: Intervention arm
Dietary Supplement: Microcrystalline maltose — Microcrystalline maltose as placebo
  Arms: Placebo arm

SUMMARY:
This trial will determine if a well-established probiotic, Vivomixx, can modulate maternal microbiota and ameliorate maternal environmental enteropathy which compromises growth in the first 1000 days. The probiotic Vivomixx has been used in many thousands of people including pregnant women, both within and outside a research context. This trial is the first in a proposed series of proof-of-concept intervention studies which are intended to provide data to enable a rational selection of interventions to be evaluated at scale in future large scale trials in which birth outcomes and postnatal growth will be key endpoints.

DETAILED DESCRIPTION:
Stunting in young children refers to attenuated linear growth. In the year 2020, 149.2 million children under the age of 5 years of age were stunted, accounting for 22% of stunting globally. Stunting has short- and long-term consequences of increased morbidity and mortality, impairment of neurocognitive development, impaired responses to oral vaccines, and increased risk of noncommunicable diseases. Stunting is partly driven by Environmental Enteric Dysfunction (EED), an enteropathic condition characterised by altered gut permeability, infiltration of immune cells and changes in villous architecture and cell differentiation. EED may help explain why nutritional supplementation either during pregnancy or early childhood has minimal value in correcting childhood stunting. Indeed, EED is believed to be responsible for 40% of childhood stunting.

Disruption in intestinal barrier function affects gut immune homeostasis, nutrient flows, and consequently dysbiosis in the gut microbiome. The gut microbiota consists of 100 trillion bacteria which interact with epithelial cells, the mucus layer and the mucosal immune system that balances tolerance and effector functions. Thus, the gut microbiome has an important role in shaping the responsiveness of the gut immune system. The mucus barrier and the normal gut microbiota limit enteropathogen colonisation. Influx of bacteria from the lumen to the systemic circulation represents microbial translocation and initiation of systemic of inflammatory process through recognition of pathogenassociated molecular patterns (PAMPs) by Pattern Recognition Receptors (PRRs) present on Antigen Presenting Cells (APCs). Three fundamental processes drive the epithelial damage which is so important in EED: infection, undernutrition, and immune dysfunction. Multiple clinical trials show that efforts to correct malnutrition through conventional therapies and improving hygiene and sanitation do not overcome growth deficits by more than about 10%. There is increasing interest in the use of probiotics which may allow pathogen decolonization, improve barrier function and restore overall gut homeostasis. Such therapies are at early stage of trials but may have potential in addressing the global burden of EED, by improving barrier function and gut pathophysiology.

Colonization of gut by enteropathogens is common in children with EED. These include ETEC, Campylobacter, Shigella and Salmonella species. Consistent data from Bangladesh and Zambia show that children with refractory stunting carry over four pathogens on average, whilst controls carry less than two. There is also clear evidence of altered composition of the microbiota in children with EED.

Probiotics may serve to overcome the problem of EED through all mechanisms of pathogenicity, by providing additional bacteria that may help in intestinal decolonization of pathogenic microorganisms (changing the microbiological niche), promoting epithelial healing, improving nutrient absorption, and restoration of an appropriate immune balance between tolerance and responsiveness.

To date the focus of research on childhood stunting has been on the young child. It is increasingly appreciated, however, that stunting often begins in utero and the focus has shifted to women's health and pregnancy. For example, the Lancet 2021 Series on maternal and child undernutrition states that "Investments to reduce undernutrition in women are important not only for women's own health but also for the health and nutrition of their children". Results from rural Bangladesh reveal poor gestational weight gain that ultimately leads to intrauterine growth restriction, low birth weight and ultimately stunting and wasting. Furthermore, another study recently completed in slum settlements of Dhaka, Bangladesh demonstrated a high prevalence of EED among undernourished women. Intestinal histopathology was abnormal in more than 80% of women. We postulate that growth retardation in utero is a consequence of EED in the mother during pregnancy and lactation. This leads to systemic inflammation, which leads to disadvantageous partitioning of nutrients, and reduced nutrient availability.

This trial will explore the conceptual framework that a well-known probiotic, that can improve the composition of the gut microbiota, can also reduce biomarkers of intestinal inflammation and gut health. This will restore healthy microbial signalling to the host epithelium, ameliorate barrier function through secretion of mucus and antimicrobial factors, and improve nutrient availability.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older in the first trimester or early second trimester of pregnancy, living in defined geographical areas of Bangladesh (Matlab), Pakistan, Senegal and Zambia, where it can be assumed that environmental enteropathy is universal

Exclusion Criteria:

* Potential participants will not be enrolled if they:

  * have had diarrhea, defined as the passage of three or more loose stools per 24 hours, in the preceding 14 days
  * have taken antibiotics or probiotics in the preceding 14 days
  * have taken steroids or non-steroidal anti-inflammatory drugs in the preceding 14 days
  * have severe pallor (hemoglobin concentration <8g/dl)
  * have any chronic disease, illness or condition which in the opinion of the investigator will complicate the assessment of safety or efficacy
  * have any gastrointestinal contraindication to ingestion of a capsule (known or suspected gastrointestinal obstruction, stricture, fistula, gastroparesis, or any swallowing disorder)
  * have the plan to observe fast at any time during the intervention period
  * have the plan to leave the study area within the follow-up period
  * are included in any other intervention trial
  * belong to a household from which another woman is already enrolled in the study

but may be enrolled if/when these disqualifiers have expired

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage change (mean, unweighted) in a multiple panel of biomarkers between baseline and last sample collected after 56 days of treatment, compared to control group | 56 days
  Plasma CRP, AGP, sCD14, LBP, CD163, iFABP, and fecal myeloperoxidase, neopterin, calprotectin and lipocalin by ELISA

SECONDARY OUTCOMES:
Reduction in colonisation | 56 days
  Specific enteropathogens (Salmonella, Shigella, Campylobacter, ETEC, EPEC, EAEC, rotavirus, norovirus, Giardia and Cryptosporidium) by TaqMan Array cards, between baseline and last sample collected after 56 days of treatment, in Vivomixx compared to placebo groups
Change in microbiome | 56 days
  Measured by whole-genome shotgun metagenomic sequencing, post versus pre intervention, in the intervention and placebo groups
Change in untargeted metabolome | 56 days
  Measured by LC-MS/MS in fecal and CapScan samples
Reduction in intestinal permeability | 56 days
  Measured by lactulose-rhamnose (LR) ratio in Vivomixx compared to placebo group
Change in weight gain velocity in the 2nd trimester of pregnancy | 14 weeks
  Rate of weight gain (kg/week)

OTHER OUTCOMES:
Recovery of useful data from CapScan | 56 days
  Completion of whole gut microbiome profiles
Diversity, centroids and distributions of microbial taxa from sequenced CapScan samples | 56 days
  microbial taxa of stool Analyzing samples from the same study population
Fetal growth | 6 months
  Using serial pregnancy ultrasound
Stillbirth | At birth
  Death or loss of a baby before or during delivery
Neonatal death | From birith to 28 days after birth
  Death of a child within 28 days after birth
Preterm birth | At birth
  Babies born alive before 37 weeks of pregnancy are completed
Apgar score | At birth
  A measure of the physical condition of a newborn infant (0-10)
Birth weight | At birth/7 days within birth
  Infant weight at birth in grams
Birth length | At birth/7 days within birth
  Infant length at birth in cm
Birth head circumference | At birth/7 days within birth
  Infant head circumference at birth in cm
Low birth weight | At birth/7 days within birth
  birth weight less than 2500 g
Small for gestational age | At birth/7 days within birth
  Birth weight of less than 10th percentile for gestational age
Women's mental health | 2 years
  By follow ups
Women's postpartum weight loss/retention | 1 year
  Follow ups
Infant weight | 1 year
  Infant weight in grams
Infant length | 1 year
  Infant length in cm
Infant morbidity | 1 year
  Number of episodes of any morbidity

CONTACTS AND LOCATIONS:
Overall Officials: S. M. Tafsir Hasan, MBBS, MS, Principal Investigator — Nutrition Research Division, icddr,b
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Chāndpur, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided